CLINICAL TRIAL: NCT06819956
Title: Ketorolac at Lower Doses for Analgesic Pain Control in ICU: A Randomized, Blinded, Parallel-Group, Placebo-Controlled Trial to Ascertain the Effect of Ketorolac on Pain Scores and Opiate Use for Critically Ill Patients
Brief Title: Ketorolac at Lower Doses for Analgesic Pain Control in ICU: A Pilot Feasibility Study
Acronym: KETOROLAC-ICU
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00126948
Record Dates: First submitted 2025-01-30; First posted 2025-02-11 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Pain Management
Keywords: analgesia; ketorolac; NSAID; ICU
MeSH Terms: conditions — Agnosia | interventions — Ketorolac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketorolac (Experimental): Ketorolac administration + standard of care.
  Participants will not be allowed to have co-administered alternative NSAIDs during the duration of their exposure on the study drug. After each administered dose, overall analgesic requirements should be assessed by the treating team (as per local institutional guidelines and practices), with attempts to wean analgesic infusions or use reduced doses of analgesic medications (especially if objective pain score measures are zero, e.g. CPOT or NRS/VAS).
  Interventions: Drug: Ketorolac
- Placebo (Placebo Comparator): Placebo administration + standard of care.
  Participants will not be allowed to have co-administered alternative NSAIDs during the duration of their exposure on the study drug. After each administered dose, overall analgesic requirements should be assessed by the treating team (as per local institutional guidelines and practices), with attempts to wean analgesic infusions or use reduced doses of analgesic medications (especially if objective pain score measures are zero, e.g. CPOT or NRS/VAS).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketorolac — Ketorolac 15 mg IV q6h for a maximum of 3 days total or discharge from ICU (whichever comes first). The ketorolac will be diluted in a 0.9% normal saline 10 mL syringe.
  Arms: Ketorolac
Drug: Placebo — Matching placebo IV q6h for a maximum of 3 days total or discharge from ICU (whichever comes first). The matching placebo will be diluted in a 0.9% normal saline 10 mL syringe.
  Arms: Placebo

SUMMARY:
Opiates are commonly used to control pain in critically ill patients in the ICU. However, increased rates of opiate use in hospital may lead to increased prescription-based opiate dependence after leaving the ICU. This may contribute to the ongoing opiate epidemic across the world. Other medications that can reduce pain, like non-steroidal anti-inflammatory drugs (NSAIDs), are being studied in critically ill patients. These drugs block the enzyme, cyclooxygenases (COX), which causes inflammation in the body. Blocking these enzymes can decrease pain, fever, and inflammation. Traditionally, NSAIDs are not commonly used in critically ill patients due to the perceived risk of gastrointestinal (GI) bleeding and acute kidney injury (AKI). However, many critically ill patients are already receiving medications and treatments to prevent GI bleeding and AKI and are closely monitored so these medications may be useful in reducing pain for these patients.

The purpose of this study is to see whether NSAIDs can be used safely in critically ill patients to reduce the dose of opiates required for pain control. This is a pilot study or a feasibility study, which is not expected to answer the question definitively. Its main purpose is to determine if NSAIDs could reduce the use of opiates in critically ill patients while in the ICU. The data collected in this study may be used in a larger study in the future.

DETAILED DESCRIPTION:
Purpose: The purpose of this study is to determine the feasibility of conducting a future, adequately powered large-scale randomized trial, while evaluating the safety and efficacy of an intravenous NSAID (e.g., ketorolac) plus usual care as compared to placebo plus usual care in critically ill patients.

Hypothesis: The investigators hypothesize that this single-centre pilot study will demonstrate that NSAIDs administration is feasible and safe in ICU patients and may potentially reduce opiate use in ICU patients with pain.

Justification: Pain control in ICU is difficult to achieve given that opiates are the mainstay of analgesia in critically ill patients, but this is not without unintended side effects, especially unintended consequences of possible future drug dependence or addictions. Given that opiates and other adjunctive pain medications (e.g., acetaminophen) are being utilized at high proportional rates, and that NSAIDs are used at relatively low rates (due to the theoretical risk of increased AKI and GI bleeds), there is potential for practice change for increased NSAID use at lower doses to reduce pain and opiate use, while not increasing risks.

Objectives: The primary objective of this pilot trial is to assess the feasibility of a larger clinical trial utilizing NSAIDs in the ICU for patients with pain. The primary outcomes of the pilot feasibility trial are: recruitment and consent rates, proportion of eligible participants who are randomized vs. not randomized, retention and protocol adherence rates.

The secondary objectives are to assess safety of the proposed trial (e.g. gastrointestinal bleeding, acute kidney injury, death) and efficacy outcomes (e.g. participant pain scores, opiate and other analgesia usage).

Research Methods/Procedures: The investigators have designed KETOROLAC-ICU as a pilot randomized controlled trial (prospective, single centre, parallel-group, concealed, blinded) examining the use of low-dose ketorolac for critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Admission to intensive care unit (ICU)
* Participants with pain (Critical Care Pain Observation Tool [CPOT] > 1 and/or self-report pains score >1 on visual analogue scale [VAS] or numerical rating scale [NRS])

Exclusion Criteria:

* Serum Cr > 100 mmol/L for females, and >130 mmol/L for males
* Ongoing ACEi (angiotensin converting enzyme inhibitor)/ARB (angiotensin receptor blocker) use in ICU
* Known hyperkalemia > 5.5
* Pre-existing chronic kidney disease (CKD Stage > 3), defined by a serum Cr > 100 mmol/L for females, and >130 mmol/L for males (at the time of screening, based on pre-hospital stable outpatient baseline values)
* New acute kidney injury KDIGO Stage > 2 (increased more than > 2-to-3 times in serum creatinine above baseline AND/OR <0.5mL/kg/hour urine output for >12 hours)
* Pre-existing gastrointestinal bleeding (within 12 weeks of hospital admission, requiring hospitalization or medical evaluation), new peptic ulcer disease, esophagitis, esophageal varices within the last 3 months
* Active gastric / duodenal / peptic ulcer, active GI bleeding
* Prior contraindications/allergies to NSAIDS or stress ulcer prophylaxis, specifically if a participant has had an anaphylactic reaction (asthma or urticaria) or non-anaphylactic asthma reaction to NSAIDs or any stress ulcer prophylaxis, e.g. proton pump inhibitor, histamine-2-blockers, etc. (e.g. proton pump inhibitor, histamine-2-blockers, etc.)
* Complete or partial syndrome of ASA-intolerance (e.g. rhinosinusitis, urticaria/angioedema, nasal polyps, asthma)
* Participants who are not receiving stress ulcer prophylaxis (e.g. proton pump inhibitor, histamine-2-blockers, etc.) while in ICU
* Any active bleeding (requiring any blood products or adjunctive coagulation agents, any output of blood >100 mL/hr, e.g. chest tube drainage, abdominal cavity drain, etc.)
* Currently receiving NSAID(s) for another indication
* Inflammatory bowel disease (e.g. participants with prior diagnosis of Crohn's disease or ulcerative colitis)
* Receiving probenecid, oxpentifylline or pentoxifylline
* Active ischemic heart disease (acute myocardial infarction, acute coronary syndrome during current hospital admission)
* Moderate-severe uncontrolled heart failure (New York Heart Association: Class II-IV)
* Moderate to severe liver impairment or active liver disease (Operational definition: participants with prior history of Child-Pugh class B (moderate) or C (severe) liver cirrhosis, OR Model for End-Stage Liver Disease-Sodium (MELD-Na) score >25, OR active acute liver failure: severe acute liver injury with encephalopathy and impaired synthetic function International Normalized Ratio (INR) >1.5 with or without pre-existing liver disease)
* Active cerebrovascular bleeding or stroke (cerebrovascular accident, transient ischemic attacks and/or amaurosis fugax, e.g. participants with active stroke symptoms within current hospital admission)
* Cerebrovascular bleeding or other bleeding disorders
* Coagulation disorders, post-operative patients with high haemorrhagic risk or incomplete haemostasis in patients with suspected or confirmed cerebrovascular bleeding
* Neuraxial (epidural or intrathecal) administration of ketorolac tromethamine injection due to its alcohol content
* Rhabdomyolysis (creatinine kinase >5000 U/L)
* Recent transplant (during same hospital admission, e.g., heart, lung, kidney, liver, etc.)
* Known allergy to ketorolac or other NSAIDs
* Participants expected to stay in ICU < 48 hours
* In the opinion of the attending physician, expected death or withdrawal of life-sustaining treatments within 48 hours
* Participant is known to be pregnant and/or breastfeeding
* Most responsible physician, participant, or substitute decision maker declines study participation (and reason)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility - Recruitment and Retention | Days 1-7, 90
  Recruitment rate at pilot site (participants/month), consent rates of eligible participants, proportion of eligible participants not randomized, and participant retention rates.
Feasibility - Protocol Adherence | Days 1-7, 90
  Rates of protocol adherence and reasons for protocol non-adherence.

SECONDARY OUTCOMES:
Opioid Use | Baseline; Days 1-7, 14, 21, 28, 90
  The administration of opioid medications (converted into oral morphine equivalents)
Pain Scores - Critical Care Pain Observation Tool (CPOT) | Baseline; Days 1-7, 14, 21, 28
  The critical care pain observation tool (CPOT) is used by healthcare workers to measure four indicators of pain: facial expression, body movements, muscle tension, and compliance with the ventilator (or vocalization for extubated participants). Each of the four indicators are ranked from 0 to 2, with higher numbers describing more pain behaviors.
Pain Scores - Visual Analog Scale (VAS) | Baseline; Days 1-7, 14, 21, 28
  The visual analog scale (VAS) is a self-reported measure of a participant's level of pain. This tool consists of a single, 10cm long line, with one end titled "No pain" and the other end titled "Pain as bad as it could possibly be." The participant then draws a mark on the line that corresponds to their level of pain. This mark is later quantified in distance from the "no pain" side of the line.
Pain Scores - Numerical Pain Rating Scale (NRS) | Baseline; Days 1-7, 14, 21, 28
  The numerical pain rating scale (NRS) is a self-reported measure of a participant's level of pain. Participants are asked to rank their pain on a scale of 0 to 10, with 0 representing no pain, and 10 representing the worst possible pain.
Safety - Acute Kidney Injury | Days 1-7, 28
  KDIGO Stage ≥ 2 (increased serum creatinine > 2-3 times above baseline AND/OR <0.5mL/kg/hour urine output for >12 hours) AND/OR need for renal replacement therapy
Safety - Gastrointestinal (GI) Bleeding | Days 1-7, 28
  Clinically significant GI bleeding (visual and physiological evidence of overt GI bleeding)
Safety - Other | Days 1-28
  Occurrence of any adverse and/or serious adverse events
All-Cause Mortality | Days 28, 90
  All-cause mortality in ICU, in hospital, or post-discharge.
Health-Related Quality of Life (EQ-5D-5L) | Day 90
  EuroQol's Health-Related Quality of Life questionnaire (EQ-5D-5L) is a self-reported measure of a participant's current health status and quality of life. This questionnaire consists of 5 questions, each representing a different dimension of health-related quality of life: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each question has 5 possible responses, ranging from "no problem" (score of 1) to "unable/extreme problems" (score of 5).
Clinical Frailty Scale (CFS) | Baseline; Day 90
  The Clinical Frailty Scale (CFS) is a tool to describe a participant's frailty and level of functioning. This scale ranges from "Very Fit" (score of 1) to "Terminally Ill" (score of 9).
Cognitive Measures | Days 1-28
  Delirium incidence (ICDSC scores ≥ 4), duration of decreased level of consciousness (LOC) due to moderate-severe sedation (RASS scores ≤ -3), duration of decreased LOC requiring intubation or ongoing mechanical ventilation (GCS < 8)
Organ Support | Days 1-7, 14, 21, 28, 90
  Use and duration of invasive mechanical ventilation (including rates of reintubation), non-invasive ventilation, renal replacement therapy, and vasopressors
Length of Admission | Day 90
  ICU length of stay, hospital length of stay, readmission episodes
Procedures | Days 1-7, 28
  Need for endoscopy (EGD or colonoscopy), angiography, and/or exploratory laparotomy
Other Analgesia | Days 1-7, 14, 21, 28, 90
  Administration of non-opioid analgesic medications

CONTACTS AND LOCATIONS:
Overall Officials: Vincent I Lau, MD MSc, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada